CLINICAL TRIAL: NCT00219596
Title: An 8-Week, Randomized, Open-Label, Parallel Group Study Comparing The Efficacy And Safety Of Xalacom With The Combination Of Unfixed Latanoprost And Timolol In Subjects With Open-Angle Glaucoma Or Ocular Hypertension
Brief Title: Xalacom And Combination Of Unfixed Latanoprost And Timolol In Subjects With Open-Angle Glaucoma Or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6641028
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2006-11

CONDITIONS: Glaucoma, Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Xalacom; Timolol

INTERVENTIONS:
Drug: Xalacom
Drug: unfixed Latanoprost and Timolol

SUMMARY:
to compare efficacy and safety of Xalacom with the combination of unfixed Latanoprost and Timolol in subjects with open-angel glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* patients with open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* closed/barely open anterior chamber angle or a history of acute angel closure glaucoma
* Ocular surgery within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate that Xalacom is as effective as uFC latanoprost and timolol at reducing IOP in subjects with open-angel glaucoma or ocular hypertension

SECONDARY OUTCOMES:
To compare the proportion of subjects reaching specified IOP levels at Week 8 To evaluate the ocular and systemic AEs across all clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- China (6):
  - Pfizer Investigational Site, Beijing, Beijing Municipality
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Shanghai, Shanghai Municipality
  - Pfizer Investigational Site, Xi’an, Shanxi
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- [Derived] Zhao JL, Ge J, Li XX, Li YM, Sheng YH, Sun NX, Sun XH, Yao K, Zhong Z; Xalacom Study Group in China. Comparative efficacy and safety of the fixed versus unfixed combination of latanoprost and timolol in Chinese patients with open-angle glaucoma or ocular hypertension. BMC Ophthalmol. 2011 Aug 19;11:23. doi: 10.1186/1471-2415-11-23. PMID 21851642